CLINICAL TRIAL: NCT04091945
Title: A Phase IIa, Double-Blind, Single Dose, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Potential Efficacy of LT3001 Drug Product in Subjects With Acute Ischemic Stroke (AIS)
Brief Title: A Study to Evaluate the Safety and Potential Efficacy of LT3001 Drug Product in Subjects With AIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lumosa Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LT3001-201
Record Dates: First submitted 2019-09-05; First posted 2019-09-17 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LT3001 Drug Product (Active Comparator)
  Interventions: Drug: LT3001 Drug Product
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LT3001 Drug Product — Active comparator
  Arms: LT3001 Drug Product
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, single-dose, randomized, and placebo-controlled prospective Phase IIa clinical study, designed to evaluate LT3001 drug product versus placebo/control in subjects with AIS.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 90 years
* NIHSS of 4 to 30
* Diagnosis of AIS within 24 hours after stroke symptoms onset

Exclusion Criteria:

* Treatement with approved drug during the current AIS
* Pre-stroke disability
* Imaging evidence of acute intracranial hemorrhage, intraparenchymal tumor, arteriovenous malformations, other central nervous system lesions that could increase bleeding risk, or aneurysm requiring treatment
* Suspected subarachnoid hemorrhage
* Seizure
* Uncontrolled hypertension
* INR >1.7 and/or abnormal aPTT or platelet count <100,000/mm3
* Blood glucose concentration <50 mg/dL or >400 mg/dL
* Lactating or pregnant subjects or those planning to become pregnant during the study
* Received anticoagulants and/or antiplatelet therapy and glycoprotein IIb/IIIa inhibitors within 48 hours
* AIS, myocardial infarction, serious head trauma or major surgery within 90 days
* Bleeding event within 21 days
* Puncture of noncompressible vessels within 7 days
* Severe hepatic, renal, and/or infectious disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - JFK Neuroscience Institute, JFK Medical Center, Edison, New Jersey
  - The Ohio State University - Wexner Medical Center, Columbus, Ohio
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Linkou Chang Gung Memorial Hospital, New Taipei City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Chao AC, Lee TH, Pettigrew LC, Hannawi Y, Huang HY, Chi NF, Chan L, Chen PL, Devlin T. Intravenous Odatroltide for Acute Ischemic Stroke Within 24 Hours of Onset: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study. Drug Des Devel Ther. 2024 Jun 6;18:2033-2042. doi: 10.2147/DDDT.S460831. eCollection 2024. PMID 38859883

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LT3001 Drug Product | Placebo
Started | 16 | 8
Completed | 14 | 7
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LT3001 Drug Product | Placebo | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (12.63) | 67.6 (9.24) | 63.9 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 12 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 3 | 18
  Unknown or Not Reported | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 5 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subject Have Symptomatic Intracranial Hemorrhage (sICH) of a Single Dose LT3001 Drug Product in Subjects With AIS.
Description: Compare the the percentage of subject having sICH between LT3001 drug product and Placebo.
Time Frame: Within 36 hours
Measure: Count of Participants; unit: Participants
Arm/Group | LT3001 Drug Product | Placebo
Number analyzed (Participants) | 16 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time the subject received the IP until the last follow-up visit, approximately 92 days.
Arm/Group | LT3001 Drug Product | Placebo
All-Cause Mortality (participants affected / at risk) | 1/16 | 1/8
Serious Adverse Events (participants affected / at risk) | 4/16 | 2/8
Other Adverse Events (participants affected / at risk) | 16/16 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LT3001 Drug Product (N=16) | Placebo (N=8)
Pneumonia (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Stroke in evolution (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LT3001 Drug Product (N=16) | Placebo (N=8)
Constipation (Gastrointestinal disorders) | 10 | 4
Headache (Nervous system disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypertension (Vascular disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Pneumonia (Infections and infestations) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Oedema peripheral (General disorders) | 2 | 1
Tachycardia (Cardiac disorders) | 2 | 0
C-reactive protein increased (Investigations) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Brain oedema (Nervous system disorders) | 3 | 0
Stroke in evolution (Nervous system disorders) | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT04091945/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT04091945/SAP_003.pdf